CLINICAL TRIAL: NCT02221934
Title: High-Frequency Nerve Block for Post-Amputation Pain: A Pivotal Study
Brief Title: Electrical Nerve Block for Amputation Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuros Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 003-0001; QUEST Trial (Other: Neuros Medical)
Record Dates: First submitted 2014-08-15; First posted 2014-08-21 (Estimated); Results first posted 2023-09-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-10

CONDITIONS: Post-Amputation Pain; Phantom Limb Pain; Residual Limb Pain; Stump Pain
Keywords: Pain; Chronic; Amputation; Phantom Pain; Stump Pain
MeSH Terms: conditions — Phantom Limb; Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test Treatment (Experimental): Self-initiated high frequency bioelectric nerve block delivered to the nerve by Altius.
  Interventions: Device: Altius
- Active Sham Control Treatment (Active Comparator): Self-initiated non-therapeutic electrical signal delivered to the nerve by Altius.
  Interventions: Device: Altius

INTERVENTIONS:
Device: Altius — Electrical signal

SUMMARY:
The purpose of the clinical trial is to learn whether electrical nerve block via the Altius System is a safe and effective treatment for patients with post-amputation pain.

DETAILED DESCRIPTION:
The Altius System is an implanted device designed to electrically block nerve signals and alleviate pain. Use of this device may be associated with providing an effective, mechanism-based yet non-destructive, treatment for managing intractable limb pain in amputees. In a given patient, the Altius System will be deemed effective if treatment results in 50% reduction of pain score for more than 50% of all pain episodes.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 21 years old
* Unilateral amputated leg ≥ 12 months
* Chronic post amputation pain ≥ 6 months
* Pain episodes typically lasting ≥ 60 minutes
* Stable drug regimen ≥ 4 weeks
* No changes to medications or prosthesis for 3-month primary study period

Key Exclusion Criteria:

* Implanted with an active implantable medical device (i.e. pacemaker)
* Confounding source of pain that interferes with reporting of limb pain
* Uncontrolled diabetes
* Spasticity preventing full range of motion of involved side
* Extremely short stump; sits on end
* Untreated psychological condition (i.e. borderline personality)
* Condition requiring MRI studies or diathermy after device implant
* Life expectancy of less than 24 months
* Progressive neurological disease (i.e. multiple sclerosis)
* Subjects with active local or systemic infection or immunocompromised

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-09-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Kapural, MD, PhD, Principal Investigator — Center for Clinical Research, Winston-Salem NC
Locations (22):
- United States (22):
  - Arizona Pain Institute, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - HCA Healthcare Research Institute / St. Luke's Presbyterian, Denver, Colorado
  - Nona Medical Arts, Orlando, Florida
  - Emory University / Grady Hospital, Atlanta, Georgia
  - Legacy Brain & Spine LLC, Atlanta, Georgia
  - Drug Studies America, Marietta, Georgia
  - University of Illinois Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic Pain Management, Cleveland, Ohio
  - Meta Medical Research Institute, Dayton, Ohio
  - Kettering Medical Center, Springboro, Ohio
  - Advanced Surgical and Research Solutions, Oklahoma City, Oklahoma
  - Cardiovascular Surgery Clinic, Memphis, Tennessee
  - The Surgical Clinic, Nashville, Tennessee
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Baylor Scott and White - Temple Memorial Vascular Surgery, Temple, Texas
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soin A, Shah NS, Fang ZP. High-frequency electrical nerve block for postamputation pain: a pilot study. Neuromodulation. 2015 Apr;18(3):197-205; discussion 205-6. doi: 10.1111/ner.12266. Epub 2015 Feb 5. PMID 25655583
- [Background] Kapural L, Syed Shah N, Fang ZP, Mekhail N. Multicenter, Double-Blinded, Randomized, Active-Sham Controlled Clinical Study Design to Assess the Safety and Effectiveness of a Novel High Frequency Electric Nerve Block System in the Treatment of Post-Amputation Pain (The QUEST Study). J Pain Res. 2022 Jun 3;15:1623-1631. doi: 10.2147/JPR.S353674. eCollection 2022. PMID 35685299
- [Result] Kapural L, Melton J, Kim B, Mehta P, Sigdel A, Bautista A, Petersen EA, Slavin KV, Eidt J, Wu J, Elshihabi S, Schwalb JM, Garrett HE Jr, Veizi E, Barolat G, Rajani RR, Rhee PC, Guirguis M, Mekhail N. Primary 3-Month Outcomes of a Double-Blind Randomized Prospective Study (The QUEST Study) Assessing Effectiveness and Safety of Novel High-Frequency Electric Nerve Block System for Treatment of Post-Amputation Pain. J Pain Res. 2024 Jun 6;17:2001-2014. doi: 10.2147/JPR.S463727. eCollection 2024. PMID 38860215
- [Result] Kapural L, Kim B, Eidt J, Petersen EA, Schwalb JM, Slavin KV, Mekhail N. Long-Term Treatment of Chronic Postamputation Pain With Bioelectric Nerve Block: Twelve-Month Results of the Randomized, Double-Blinded, Cross-Over QUEST Study. Neuromodulation. 2024 Dec;27(8):1383-1392. doi: 10.1016/j.neurom.2024.08.010. Epub 2024 Sep 24. PMID 39320284
- See also: Neuros HFNB Pilot Study - Abstract — https://www.ncbi.nlm.nih.gov/pubmed/25655583
- See also: QUEST 3-month (Primary) RCT Outcomes — http://www.ncbi.nlm.nih.gov/pubmed/38860215
- See also: QUEST 12-month (Secondary) Long Term Outcomes — http://www.ncbi.nlm.nih.gov/pubmed/39320284
- See also: QUEST Study Design — http://www.ncbi.nlm.nih.gov/pubmed/35685299

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were required to fulfill all eligibility requirements, including lidocaine injection screening. Eligible subjects underwent study device implant and activation prior to group assignment.
Groups:
- Not Yet Randomized: Not yet randomized to Test Treatment or Active Sham Control Treatment groups.
Period: Screening
Arm/Group | Test Treatment | Active Sham Control Treatment | Not Yet Randomized
Started | 0 | 0 | 607
Completed | 0 | 0 | 183
Not Completed | 0 | 0 | 424
Period: Device Activation
Arm/Group | Test Treatment | Active Sham Control Treatment | Not Yet Randomized
Started | 0 | 0 | 183
Primary Safety Analysis Cohort | 0 | 0 | 183
Successful Implant | 0 | 0 | 180
Completed | 0 | 0 | 178 (178 Subjects were implanted with the study device and randomized.)
Not Completed | 0 | 0 | 5
Period: Randomized Testing (Month 1 to Month 3)
Arm/Group | Test Treatment | Active Sham Control Treatment | Not Yet Randomized
Started | 87 | 91 | 0
Successful Randomization | 87 | 91 | 0
Successful Device Use (Primary Effectiveness Analysis Cohort) | 85 | 85 | 0
Completed | 82 | 83 | 0
Not Completed | 5 | 8 | 0
Period: Follow-up (Month 3 to Month 12)
Arm/Group | Test Treatment | Active Sham Control Treatment | Not Yet Randomized
Started | 82 | 83 | 0
Completed | 74 | 75 | 0
Not Completed | 8 | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Treatment | Active Sham Control Treatment | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.21) | 57.9 (12.57) | 58.0 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 51 | 51 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 83 | 84 | 167
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 10 | 22
  White | 66 | 71 | 137
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 2 | 4
Level of Amputation [Count of Participants; unit: Participants]
  Above knee (AKA) | 38 | 35 | 73
  Below knee (BKA) | 47 | 50 | 97

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint: Reduction of Pain Level by 50% From Baseline
Description: Demonstration of 50% reduction in a Numerical Rating Scale (NRS; 0-10 Scale; with 10 being the highest pain imaginable) pain score from pre-treatment to post-treatment for more than 50% of all pain episodes. Study success will be determined by a superiority test on the difference between responder rates in the Test group (those receiving the treatment) and Control group (those who do not receive treatment).
Time Frame: Randomized Testing Window (Month-1 to Month-3 post implant, 2 Month duration)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Treatment | Active Sham Control Treatment
Number analyzed (Participants) | 85 | 85
Participants | 21 | 6
Statistical Analysis 1: Comparison: Test Treatment vs Active Sham Control Treatment; Test type: Superiority; p = 0.002, Regression, Logistic; Risk Difference (RD) = 0.176, 95% CI 2-sided [0.070 to 0.283] — Difference in Responders between groups presented

2. Primary Outcome: Primary Safety Endpoint: Incidence of Reported and Adjudicated Serious Adverse Events
Description: Incidence of all serious adverse events including serious adverse device events and unanticipated adverse device events.
Time Frame: From screening injection visit through 3 months post implant
Measure: Count of Participants; unit: Participants
Arm/Group | Test Treatment | Active Sham Control Treatment
Number analyzed (Participants) | 85 | 85
Participants
  All Serious Adverse Events (SAE) | 24 | 19
  Serious Adverse Device Effect (SADE) | 3 | 5
  Unanticipated Adverse Device Effect (UADE) | 0 | 0

3. Secondary Outcome: Secondary Effectiveness: Pain Relief After 2 Hours
Description: Average percent change of pain intensity from before treatment, 30 minutes post treatment, and 2 hours post treatment
Time Frame: 12 months post implant
Reporting Status: Not Posted

4. Secondary Outcome: Secondary Effectiveness: Pain Medication Use
Description: Average morphine equivalent dose per day over two weeks compared at Month 3, Month 6 and Month 12 to Baseline.
Time Frame: 12 months post implant
Reporting Status: Not Posted

5. Secondary Outcome: Secondary Effectiveness: Pain Interference to Activities of Daily Living (ADL
Description: Brief Pain Inventory summary score compared at Month 3, Month 6 and Month 12 to Baseline.
Time Frame: 12 months post implant
Reporting Status: Not Posted

6. Secondary Outcome: Secondary Effectiveness: Health-related Quality of Life (HR-QOL)
Description: EQ-5D summary index, SF-12 physical component and mental component summary compared at Month 3, Month 6 and Month 12 to Baseline.
Time Frame: 12 months post implant
Reporting Status: Not Posted

7. Secondary Outcome: Secondary Effectiveness: Patient Global Impression of Change (PGIC)
Description: Comparison of Patient Global Impression of Change across the Month 3, Month 6 and Month 12 office visits
Time Frame: 12 months post implant
Reporting Status: Not Posted

8. Secondary Outcome: Secondary Safety
Description: Incidence of all Non-Serious Adverse Events, including Non-Serious Adverse Events, Non-Serious Adverse Device Events, and Unanticipated (Non-Serious) Adverse Device Events from the time of consent through 12 months post implant.
Time Frame: 12 months post implant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From time of lidocaine injection screening through Month-12, approximately 1 year
Arm/Group | Test Treatment | Active Sham Control Treatment
All-Cause Mortality (participants affected / at risk) | 1/85 | 2/85
Serious Adverse Events (participants affected / at risk) | 35/85 | 35/85
Other Adverse Events (participants affected / at risk) | 34/85 | 34/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Treatment (N=85) | Active Sham Control Treatment (N=85)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Implant site necrosis (General disorders) | 0 (0) | 1 (1)
Medical device discomfort (General disorders) | 4 (4) | 1 (1)
Medical device site discomfort (General disorders) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 1 (1) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 3 (4) | 1 (1)
Incision site abscess (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4)
Postoperative wound infection (Infections and infestations) | 2 (3) | 3 (3)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Shunt infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Calcifying fibrous pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amputation stump pain (Nervous system disorders) | 2 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Device extrusion (Product Issues) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Treatment (N=85) | Active Sham Control Treatment (N=85)
Medical device discomfort (General disorders) | 5 (5) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 19 (38) | 18 (28)
Corona virus infection (Infections and infestations) | 4 (4) | 5 (5)
Postoperative wound infection (Infections and infestations) | 1 (1) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
A single-cross-over design (and not double-- cross-over) prohibited further evaluation of duration of therapy effectiveness after removal of therapy. While interesting, this would not have been in the best interests of the trial patients who required therapy to treat their chronic amputation pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT02221934/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT02221934/SAP_001.pdf